CLINICAL TRIAL: NCT01237470
Title: The Desarda and Lichtenstein Techniques in Primary Hernia Treatment in Adult Males: Randomised, Multicenter, Blinded Study.
Brief Title: The Desarda and Lichtenstein Techniques in Inguinal Hernia Treatment.
Acronym: DESLICH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: protocol completed
Sponsor: Nicolaus Copernicus University (Other)
Responsible Party: Nicolaus Copernicus University, Nicolaus Copernicus University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Nicolaus Copernicus University
Record Dates: First submitted 2010-11-08; First posted 2010-11-09 (Estimated); Last update posted 2010-11-09 (Estimated); Status verified 2010-07

CONDITIONS: Hernia, Inguinal
Keywords: inguinal hernia; hernia recurrence; no mesh techniques; Desarda technique
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Desarda group (Experimental): Patients with primary inguinal hernia operated using the Desarda technique
  Interventions: Procedure: Desarda technique
- Lichtenstein group (Experimental): Patients with primary inguinal hernia operated using the Lichtenstein technique.
  Interventions: Procedure: Lichtenstein technique

INTERVENTIONS:
Procedure: Desarda technique — no mesh technique with undetached strip of external oblique aponeurosis placed at the floor of inguinal canal
  Arms: Desarda group
Procedure: Lichtenstein technique — hernioplasty with the usage of plain polypropylene mesh
  Other Names: open plain mesh technique
  Arms: Lichtenstein group

SUMMARY:
Contemporary treatment of inguinal hernia is generally based on surgical methods with the use of synthetic meshes. The implanted meshes however have some disadvantages: they increase the risk of infection, tend to sustain inflammation process, can generate chronic pain and fertility disorders, can move from the initial implantation site, increase costs of treatment etc. The research to find any new hernioplasty without the use of meshes is still going on.

Desarda in 2002 year published his own results over hernia treatment with the use of external oblique aponeurosis. These results were comparable with the effects of Lichtenstein technique.

The initial assessment done in our own department revealed good clinical results after hernia treatment with Desarda's method.

To make appropriate and objective clinical assessment of the Desarda's technique for primary inguinal hernia treatment the randomized multicentre double blinded clinical trial (RCT) was projected and conducted. Finally, 105 patients were included in the Desarda group and 103 in the Lichtenstein group. Personal clinical follow up was made up to 3 years after operation.

Generally no statistically significant differences were found between these groups. The only difference was higher rate of seroma after Lichtenstein technique and different pain perception in both groups. To the summary it is clear that Desarda technique is quite attractive and good proposition for operative hernia treatment without mesh. The RCT was done with the use of SharePoint Portal Server (Microsoft) which seems to be appropriate for clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* primary inguinal hernia
* male adults
* signed informed consent
* god condition of external oblique aponeurosis (assessed during the operation)

Exclusion Criteria:

* age < 18
* recurrent hernia
* incarcerated hernia
* diagnosed mental disorder
* manual reduction of hernia on inpatient
* infection at groin area
* wound or scar at the groin
* no consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2009 (Actual)
Dates: Start 2005-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
recurrence | 3 years
  hernia recurrence after surgical treatement
chronic pain | 6 months
  persistent chronic pain (lasting longer then 6 months)

SECONDARY OUTCOMES:
surgical complications | 3 years
  edema, hematoma, ecchymosis, infaction of the wound

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw Dabrowiecki, MD, PhD, Study Chair — Department of General and Endocrine Surgery, Collegium Medicum, Nicolaus Copernicus University Bydgoszcz, Poland
Locations (1):
- Department of General and Endocrine Surgery, Collegium Medicum, Nicolaus Copernicus University, Bydgoszcz, Poland

REFERENCES:
- [Background] Desarda MP. Inguinal herniorrhaphy with an undetached strip of external oblique aponeurosis: a new approach used in 400 patients. Eur J Surg. 2001 Jun;167(6):443-8. doi: 10.1080/110241501750243798. PMID 11471669
- [Background] Desarda MP. Surgical physiology of inguinal hernia repair--a study of 200 cases. BMC Surg. 2003 Apr 16;3:2. doi: 10.1186/1471-2482-3-2. PMID 12697071